CLINICAL TRIAL: NCT00525421
Title: A Randomized, Placebo-Controlled, Double-Blind Trial of a Two Week Course of Curcuminoids in Oral Lichen Planus
Brief Title: A Clinical Study of Curcuminoids in the Treatment of Oral Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nita Chainani Wu (Other)
Responsible Party: Sponsor-Investigator, Nita Chainani Wu, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H1113-30233-01
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Oral Lichen Planus
Keywords: curcuminoids; oral lichen planus; c reactive protein; interleukin 6
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Diarylheptanoids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curcumin (Experimental): Curcumin C3 Complex
  Interventions: Drug: Curcuminoids
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcuminoids — Curcuminoids tablets 2000mg three times per day for 12 days
  Other Names: Curcumin C3 Complex
  Arms: Curcumin
Drug: Placebo
  Arms: Placebo

SUMMARY:
A phase 2 randomized, placebo-controlled, double-blind trial of a two week course of curcuminoids in oral lichen planus will be conducted. 26 consecutive, eligible patients with OLP presenting to the oral medicine clinic at the University of California, San Francisco, will be enrolled. Study subjects will be randomized to receive either placebo or curcuminoids 6000mg/day for 2 weeks in three divided doses of 2000mg three times/day. Measurement of signs, symptoms, periodontal status and blood tests including complete blood count, liver enzymes, serum c reactive protein and serum interleukin-6 levels will be done at baseline and at the end of 2 weeks. A side-effects questionnaire will be administered at the 2-week follow-up.

The Numeric Rating Scale (NRS) will be used to measure symptoms and the Modified Oral Mucositis Index (MOMI) to measure clinical signs of OLP. Primary outcome is change in symptoms from baseline. Secondary outcomes are change in clinical signs, occurrence of side-effects, change in serum C-reactive protein and serum interleukin-6 levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the UCSF oral medicine clinic diagnosed with either the atrophic or the erosive form of oral lichen planus
* Study subjects must have a symptom score between 3 to 8 at the time of entry into the study. (Range of scale: zero to ten with zero being no symptoms and ten being the worst imaginable symptoms.
* Study subjects will have discontinued systemic and/or topical steroids and/or curcuminoids for at least 2 weeks before entry into the study.

Exclusion Criteria:

* Pregnancy, lactation or unwillingness to use an effective method of contraception. An attempt will be made to ascertain the date of the last menstrual period among eligible pre-menopausal women. If pregnancy cannot be ruled out, a pregnancy test will be provided to the women before enrollment into the study. - Patients younger than 21 years of age.
* Patients who cannot return for a follow-up visit at two weeks after enrollment.
* Patients who have a medical contraindication to discontinuation of systemic steroids eg. those on long term corticosteroid therapy. - Patients with a history of gastro-esophageal reflux disease, gastric / duodenal ulcers, or gallstones.
* Patients with elevated liver enzymes;
* Patients on anticoagulants or antiplatelet medications.
* Patients undergoing orthodontic treatment.
* Patients who don't read, speak or understand English.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nita Chainani-Wu, DMD, MS, PhD, Principal Investigator — University of California, San Francisco; Sol Jr. Silverman, MA, DDS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Chainani-Wu N. Safety and anti-inflammatory activity of curcumin: a component of tumeric (Curcuma longa). J Altern Complement Med. 2003 Feb;9(1):161-8. doi: 10.1089/107555303321223035. PMID 12676044
- [Background] Chainani-Wu N, Silverman S Jr, Reingold A, Bostrom A, Mc Culloch C, Lozada-Nur F, Weintraub J. A randomized, placebo-controlled, double-blind clinical trial of curcuminoids in oral lichen planus. Phytomedicine. 2007 Aug;14(7-8):437-46. doi: 10.1016/j.phymed.2007.05.003. Epub 2007 Jul 2. PMID 17604143
- [Result] Chainani-Wu N, Madden E, Lozada-Nur F, Silverman S Jr. High-dose curcuminoids are efficacious in the reduction in symptoms and signs of oral lichen planus. J Am Acad Dermatol. 2012 May;66(5):752-60. doi: 10.1016/j.jaad.2011.04.022. Epub 2011 Sep 9. PMID 21907450

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 patients with symptomatic oral lichen planus (OLP) presenting to the oral medicine clinic at the University of California, San Francisco (UCSF) between October 2007 and November 2008 were screening for this study.
Pre-assignment Details: 3 patients had elevated liver enzymes at baseline and were excluded prior to randomization
Groups:
- Curcuminoid: Curcuminoids : Curcuminoids tablets 2000mg three times per day for 12 days
- Placebo: Placebo : identical placebo tablets three times per day for 12 days
Period: Overall Study
Arm/Group | Curcuminoid | Placebo
Started | 10 (Enrollment started october 2007) | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcuminoid | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.7) | 60.8 (8.6) | 58.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Symptom Score for OLP [Number; unit: Participants] — Numerical Rating Scale (NRS): 0=No oral discomfort, 10=worst imaginable oral discomfort
  Participants
    NRS 3-5 | 5 | 6 | 11
    NRS 5.5-8 | 5 | 4 | 9
Presence of Oral Ulcerations [Number; unit: Participants]
  Ulcerations at Baseline | 3 | 4 | 7
  No Ulcerations at Baseline | 7 | 6 | 13
Past medication for OLP [Number; unit: Participants] — Subjects who used medications in the past for OLP
  Participants
    Topical Steroids | 8 | 7 | 15
    No Topical Steroids | 2 | 3 | 5
    Prednisone | 6 | 5 | 11
    No Prednisone | 4 | 5 | 9
    Azathioprine | 1 | 1 | 2
    No Azathioprine | 9 | 9 | 18
    Any Prior Medication for OLP | 9 | 8 | 17
    No Prior Medication for OLP | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Two Weeks in Symptoms and Signs of Oral Lichen Planus (OLP)
Description: Numeric Rating Scale (NRS) is patient-reported numerical score for intensity of symptoms (range 0-10, where 0=no oral discomfort and 10=worst imaginable oral discomfort; symptom score over the last 1 week was recorded at baseline, and symptom score since baseline was recorded at follow-up. For Modified Oral Mucositis Index (MOMI) each of 16 oral sites is scored by an examiner for both erythema intensity (range 0-3 where 0=normal, 1=mild, 2=moderate, 3=severe) and area of ulceration (range 0-3 where 0=none, 1=>0-0.25 cm^2, 2= >0.25-1 cm^2, 3=>=1cm^2): right (R) and left (L) buccal mucosa, labial mucosa (upper and lower), lateral tongue (R and L), dorsum of tongue (R and L), ventral tongue and floor of mouth (R and L), maxillary gingiva (R and L), mandibular gingiva (R and L), and soft and hard palate. Total score for clinical signs (MOMI) is the sum of scores for 16 sites; separate scores for erythema and ulceration are the sums of respective scores.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Placebo: Placebo: Identical placebo tablets three times per day for 12 days
Arm/Group | Curcuminoid | Placebo
Number analyzed (Participants) | 10 | 10
percent change
  NRS | -22 [-33 to -14] | 0 [-29 to 16.7]
  Erythema | -17 [-29 to -8.3] | 0 [-10 to 16.7]
  Ulceration | -14 [-60 to 0] | 0 [0 to 26.7]
  MOMI | -24 [-38 to -11] | -3.2 [-13 to 9.09]

2. Secondary Outcome: Change in Serum C-reactive Protein and Serum Interleukin-6 Levels
Description: Percentage changes from baseline to two weeks in C-Reactive protein (CLP) and interleukin-6 (IL-6).
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Curcuminoid | Placebo
Number analyzed (Participants) | 10 | 10
Percent change
  CRP | 0 [-21 to 19] | 33.3 [0 to 50]
  IL-6 | 20.3 [-16 to 60.6] | -1.6 [-6.1 to 3.17]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Side effects were recorded using a 10-item questionnaire, complete blood cell count, and measurement of liver enzymes, aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase at the 2-week follow-up visit
Arm/Group | Curcuminoid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curcuminoid (N=10) | Placebo (N=10)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated liver enzymes (Hepatobiliary disorders) | 2 (2) | 0 (0) — Liver enzymes (AST, ALT and alkaline phosphatase) assessed for change from normal baseline to abnormal at follow-up. ALT changed form 40 to 44, and from 59 to 64.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes